CLINICAL TRIAL: NCT00875342
Title: D-cycloserine Enhanced Imaginal ExposureTherapy for Posttraumatic Stress Disorder (PTSD)
Brief Title: Imaginal Exposure & D-Cycloserine (DCS) for Posttraumatic Stress Disorder (PTSD)
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Trial is no longer enrolling due to priority of other non-pharmacologic PTSD trials.
Sponsor: Weill Medical College of Cornell University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 0802009646
Record Dates: First submitted 2009-04-02; First posted 2009-04-03 (Estimated); Results first posted 2021-08-16 (Actual); Last update posted 2021-08-16 (Actual); Status verified 2021-07

CONDITIONS: Posttraumatic Stress Disorder
Keywords: Traumatic Event; Trauma Survivor; Exposure Therapy; PTSD DCS; Telemedicine; Telepsychiatry; Telemental health
MeSH Terms: conditions — Stress Disorders, Post-Traumatic

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- D-cycloserine (Experimental): 100 mg on days of therapy session
  Interventions: Drug: DCS
- Placebo (Placebo Comparator): Sugar pill
  Interventions: Other: Placebo

INTERVENTIONS:
Drug: DCS — 1. Cognitive behavioral treatment with exposure therapy plus D-Cycloserine (100 mg on days of therapy session (approximately 9 times)
  Arms: D-cycloserine
Other: Placebo — 2. Cognitive behavioral treatment with exposure therapy plus a placebo(sugar pill) (Placebo given on days of therapy session (9 times)
  Arms: Placebo

SUMMARY:
This study proposes to evaluate the effects of D-cycloserine (DCS) combined with cognitive-behavioral treatment with exposure therapy in a sample of patients who developed posttraumatic stress disorder (PTSD) as a consequence of various traumas (e.g., motor vehicle and accidents, burns and other injuries, combat, World Trade Center attack, etc.). In addition, this study hopes to determine whether a common human genetic single nucleotide polymorphism (SNP) in a growth factor, brain derived neurotrophic factor, BDNF SNP (Val66Met), predicts treatment response to PTSD.

Patients living in areas that are not geographically proximal to the Weill-Cornell Medical Center New York City campus will receive cognitive behavioral therapy using telemedicine (videoconferencing technology).

Overall, this study aims 1) to determine if subjects administered DCS show a significantly larger decrease in symptoms of PTSD as compared to those administered a placebo, 2) to determine if subjects administered DCS show a decrease in PTSD symptomatology significantly earlier (as measured by weeks) than those administered a placebo, 3) to determine if differences in symptomatology are evident at a 6-month follow-up and indicate long-term differences between groups, 4) to determine if the BDNF SNP predicts treatment response, 5)to determine if it is feasible and acceptable to provide imaginal exposure (IE) therapy for PTSD using videoconferencing technology.

DETAILED DESCRIPTION:
Following an initial assessment evaluating eligibility for the study, eligible participants will be randomly assigned to one of two treatment groups: imaginal exposure (IE) plus DCS (100mg) or IE plus placebo (sugar pill). DCS is a broad spectrum antibiotic that has recently been implicated as a cognitive enhancer and may enhance the treatment that occurs. The participant, assessor and treating clinicians will be blinded to which pill the participant is receiving. The dose of medication will need to be taken only on the days of therapy sessions during which the exposure occurs (approximately 9 times). Both groups will be treated with a standardized cognitive-behavioral exposure therapy protocol utilizing gold-standard treatment, consisting of 12-14 weekly individual (one-on-one) sessions with a highly qualified clinical psychologist. Treatment interventions include imaginal exposure, graduated in vivo exposure, psycho-education, relaxation training, behavioral activation, and cognitive restructuring. Assessments will occur prior to treatment, following sessions 3, 6 and 10, following completion of treatment, and 6 months after the conclusion of treatment. In addition, all participants will be genotyped once for the BDNF SNP (Val66Met) using a non-invasive saliva sample.

ELIGIBILITY:
Inclusion Criteria:

1. English-speaking adults
2. Age 18-70
3. Survivor of a variety of traumas (e.g., motor vehicle and accidents, burns and others injuries, combat, World Trade Center attack, etc.)
4. Diagnosed with PTSD
5. In good health. For persons with chronic injuries/conditions related to their accidents, "good health" is defined as the injury being in a state of stabilization and able to attend weekly outpatient sessions.

Exclusion Criteria:

1. Current organic mental disorder
2. Schizophrenia or symptoms of psychosis/delusions
3. Bipolar disorder
4. Current substance abuse or dependence
5. Active suicidal/homicidal ideation, intent, or plan
6. Use of pacemaker
7. Significant health impairment, including renal disease
8. Taking oral anticoagulant medication, ethionamide (Trecator-SC), isoniazid (INH), or anti-depressant medication
9. Hypersensitivity to cycloserine
10. History of seizures
11. Pregnant or currently trying to conceive, or breastfeeding

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 41 (Actual)
Dates: Start 2008-05 (Actual); Primary Completion 2018-02-28 (Actual); Study Completion 2018-02-28 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: JoAnn Difede, PhD, Principal Investigator — Weill Medical College of Cornell University
Locations (1):
- Weill Cornell Medical College, New York, New York, United States

REFERENCES:
- See also: Related Info — http://www.patss.com

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | D-cycloserine | Placebo
Started | 20 | 21
Completed | 16 | 16
Not Completed | 4 | 5

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | D-cycloserine | Placebo | Total
Number analyzed (Participants) | 20 | 21 | 41
Age, Continuous [Mean (Standard Deviation); unit: years] | 44.50 (11.75) | 40.71 (9.83) | 42.56 (10.84)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 8 | 12 | 20
  Male | 12 | 9 | 21
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  White | 14 | 16 | 30
  Black | 2 | 2 | 4
  Hispanic | 4 | 1 | 5
  Asian | 0 | 1 | 1
  Other | 0 | 1 | 1
CAPS [Mean (Standard Deviation); unit: units on a scale] — Clinician Administered PTSD Scale (CAPS). Total CAPS severity score range is 0-136. Higher values represent a worse outcome (i.e. greater severity of posttraumatic symptoms).
  units on a scale | 97.20 (17.36) | 97.43 (17.37) | 97.31 (17.15)

OUTCOME MEASURES:

1. Primary Outcome: Symptoms of Posttraumatic Stress Disorder-Clinician Administered PTSD Scale (CAPS)
Description: Clinician Administered PTSD Scale (CAPS). Total CAPS severity score range is 0-136. Higher values represent a worse outcome (i.e. greater severity of posttraumatic symptoms).
Time Frame: Immediately after the intervention, an average of 6 months
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | D-cycloserine | Placebo
Number analyzed (Participants) | 13 | 14
units on a scale | 32.31 (32.31) | 26.93 (25.06)

ADVERSE EVENTS:
Time Frame: 14 weeks
Arm/Group | D-cycloserine | Placebo
All-Cause Mortality (participants affected / at risk) | 0/20 | 0/21
Serious Adverse Events (participants affected / at risk) | 0/20 | 0/21
Other Adverse Events (participants affected / at risk) | 0/20 | 0/21

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2009-12-11): https://cdn.clinicaltrials.gov/large-docs/42/NCT00875342/Prot_SAP_000.pdf